CLINICAL TRIAL: NCT03144466
Title: Phase I Study of the Anti-PD1 Immune Checkpoint Inhibitor Pembrolizumab And Platinum in Combination With Radical radiotherApY in Cervix cAncer.
Brief Title: A Study of Pembrolizumab And Platinum With Radiotherapy in Cervix Cancer
Acronym: PAPAYA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment.
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4268
Record Dates: First submitted 2017-04-12; First posted 2017-05-08 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2018-10

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A - Starting dose (Experimental): 100mg of pembrolizumab in n=3 patients, administered in 8 cycles every 3 weeks for a total of 18 weeks commencing two weeks prior to first fraction of radiotherapy and given in combination with Radical Radiotherapy, Brachytherapy and Cisplatin Chemotherapy. Increase in cohort by three patients to n=6 patients provided no more than 1/3 patients experience a Dose Limiting Toxicity (DLT).
  Interventions: Combination Product: Pembrolizumab
- Part A - Escalation dose (Experimental): Escalation of dose to 200mg of pembrolizumab in a further n=3 patients provided no more than 1/6 patients at starting dose experience a DLT. Increase in cohort by three patients to n=6 patients provided no more than 1/3 patients experience a Dose Limiting Toxicity (DLT).
  Interventions: Combination Product: Pembrolizumab
- Part B - Expansion phase (Experimental): Recruitment of expansion cohort of n=14 patients using Maximum Tolerated Dose (MTD) of Pembrolizumab as determined in the dose escalation phase. MTD to be administered in 8 cycles every 3 weeks for a total of 18 weeks commencing two weeks prior to first fraction of radiotherapy and given in combination with Radical Radiotherapy, Brachytherapy and Cisplatin Chemotherapy.
  Interventions: Combination Product: Pembrolizumab

INTERVENTIONS:
Combination Product: Pembrolizumab — antiPD1 monoclonal antibody
  Other Names: KEYTRUDA

SUMMARY:
Locally advanced cervix cancers (stage 1B-IV) are usually treated with radiotherapy, concomitant cisplatin chemotherapy and brachytherapy. Failure to achieve locoregional control (LRC) remains a problem, especially in the setting of stage III/IV disease. More importantly, however, the dominant unresolved problem remains the occurrence of distant metastatic relapse. With the knowledge that 99% of all cervix cancer is associated with human papillomavirus (HPV) infection, there is a strong rationale to consider immunomodulatory strategies in the radical management of this disease. Therefore, in this research protocol the investigator will treat patients with stage 1B-IVA carcinoma of the cervix planned to receive radical radiotherapy with concomitant cisplatin and brachytherapy. The research involves adding a new therapy in the form of an antiPD1 monoclonal antibody (pembrolizumab) to the standard treatment of radiotherapy combined with cisplatin chemotherapy and brachytherapy. This treatment seeks to activate the patient's own immune system to attack the cancer cells - and the investigator believes that adding this treatment during standard treatment may be particularly effective. Patients will receive an initial dose of pembrolizumab 2 weeks before starting a course of chemoradiotherapy and brachytherapy. In the first instance, patients will receive 100 mg of pembrolizumab and, if this is safe and tolerable in the first 3 patients, the dose will be increased to 200 mg for all other patients. Radiation will be delivered on 28 occasions with chemotherapy given intravenously in weeks 0, 1, 2 and 3. Brachytherapy will be given on 3 occasions after completion of the radiation. Additional doses of pembrolizumab will be given every 3 weeks for a further 7 doses. The investigator will assess the feasibility and safety of the combination of pembrolizumab with radiotherapy and cisplatin.

DETAILED DESCRIPTION:
The study is designed to determine the safest dosage of pembrolizumab to be given in combination with chemoradiotherapy and brachytherapy for patients with locally advanced cervix cancer. The study will be run at the Royal Marsden Hospital only and is open label so both patient and doctor will know what treatment patients are receiving. Patients will receive pembrolizumab in combination with chemoradiotherapy and brachytherapy. Patients will be tested against 2 dose escalation levels (Dose Level 1/2). An initial dose of 100mg of pembrolizumab will be implemented. If dose limiting toxicity is not observed at this dose, pembrolizumab will be escalated to 200mg. A minimum of 3 patients will be required at each dose level. A minimum gap of 1 week should be left between the recruitment of the first and second patient in a new dosing level to mitigate against multiple patients suffering from any acute toxicity.

* If no dose limiting toxicity is observed at a dose level, pembrolizumab will be escalated to the next dosing level.
* If 1 in 3patients experience a dose limiting toxicity then the cohort will be expanded to 6 patients.
* If 1 in 6 patients experience a DLT then the dose will be escalated to the next dosing level.
* However if ≥ 2 in 6 patients experience a DLT then the maximum administered dose (MAD)will have been reached and the previous dosing level should be used for the expansion phase. If the MAD is reached at dose level 1 the combination therapy of pembrolizumab, cisplatin and radiotherapy will not be considered possible and the trial discontinued. Once the MTD has been determined the trial enters the expansion cohort whereby a further 14 patients are treated with the determined dosage of pembrolizumab in combination with radiotherapy, brachytherapy and cisplatin. For this study the dose limiting toxicities will be assessed by the presence of:
* >=Grade 3 gastrointestinal toxicity

  o Excluding grade 3 toxicity which resolves to grade 2 within 48 hours of medical management
* Haematological toxicity including:

  * Grade 3 thrombocytopenia with bleeding
  * Grade 4 thrombocytopenia
  * Grade 4 neutropenia lasting >7 days in the absence of growth factor support
  * Grade 4 neutropenia of any duration accompanied by fever ≥ 38.5°C and/or systemic infection
  * Any other grade ≥4 haematological toxicity
* Immune system toxicity

  * Grade 4 immune toxicity requiring treatment with corticosteroids
  * Grade 3 immune toxicity requiring corticosteroid treatment (greater than 10 mg/day prednisone or equivalent dose) for greater than 12 weeks. (For patients requiring corticosteroids at week 12 toxicity assessment, the observation period will be continued to monitor for this DLT)
* Radiotherapy treatment interruption > 5 days or failure to complete external beam radiotherapy and brachytherapy due to toxicity
* any other ≥Grade 3 non-hematologic toxicity (except nausea and vomiting) which in the opinion of the investigator is considered dose-limiting.

Escalation to the next dose level will not proceed until the following criteria are satisfied:

* If 0/3 patients experience a DLT escalation to the next dose level can proceed.
* If 1/3 patients experiences a DLT a further 3 patients will be recruited at the dose level.

  * If 1/6 patients experience a DLT then escalation to the next dose level can proceed.
  * If ≥ 2/6 patients in a specific dose level experience a DLT, the maximum tolerated dose will have been reached and all patients in the expansion cohort will be recruited at the previous dose level.
* If 2/3patients experience a DLT then the maximum tolerated dose will have been reached and the expansion cohort phase will begin at the previous dose level. If the MAD occurs at dose level 1 the expansion cohort will not go ahead and the trial will be stopped.

Patient Pathway through the Study: Once the patient consents to taking part on the trial the patient will enter the screening period. This can last from 1 to 14 days before the proposed start of the study treatment. As part of the screening period the patient will be required to attend a clinic where a doctor will complete a physical examination, assess the patients' vital signs and performance status, measure the patients' weight and collect information on the patients' medical history and any medications the patient is currently taking. Patients will also be asked to undertake routine blood tests and a MRI/PET-CT scan; if these have been completed as part of routine care; prior to consent and within the screening time lines; the results can be used for the study. Female patients will be asked to complete a pregnancy test up to 72 hours before confirmation of study eligibility. If the patient is confirmed as eligible then the patient will be receive a preloading dose of pembrolizumab (at the dosage currently under evaluation) 2 weeks prior to the start of chemoradiotherapy and then every 3 weeks until the patients have completed all 7 cycles, the patient disease progresses, the patient suffers from too many side effects or the patient decides they no longer wish to take part in the study. Whilst on treatment at each clinic visit before the drug is given the patient will also be required to attend a clinic so the doctor can complete a physical examination, assess the patients' vital signs and performance status, measure the patients' weight and collect information on any side effects the patient may have and any medications the patient is taking. At this visit the patient may also be required to give blood for routine blood tests and research blood samples if the patient have consented to do this. Once all the above assessments have been verified by the doctor Pembrolizumab will be given by a drip into the patients' arm that will take approximately 30 minutes. Patients will also be asked to attend a visit for a MRI/PET-CT at pre-brachytherapy (week 5), after the last dose of pembrolizumab (week 18) and then every 3 months for 2 years or until disease progression, discontinuation or initiation of another anticancer treatment. This is to see what is happening to the cancer as the patient continues on the study. FollowUp: When a patient completes their last dose of pembrolizumab the patient will be asked to attend post treatment follow up visit 4 weeks after their last dose of pembrolizumab and a safety follow up at 19 weeks from their last dose or before the initiation of a new anti-cancer therapy; whichever comes first. At the post treatment follow up visit and SFU visit the doctor will complete a physical examination, assess the patient vital signs and performance status, measure the patient weight and collect information on the patients' cancer, any side effects the patient may have and any medications the patient is taking. Patients will also have routine bloods taken. If the patient has completed all 8 doses and has not progressed at the safety follow-up (SFU) the patient will be reviewed for tumour progression and initiation of new anti-cancer treatments every 12 weeks for 2 years to review the disease status and if the patients have received any additional anticancer treatments until progression, initiation of a new anti-cancer therapy, withdrawal or completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed FIGO stage 1B - IVA carcinoma of the cervix planned to receive radical radiotherapy with concomitant cisplatin and brachytherapy. Pelvic lymph node but not para-aortic lymph node involvement is permitted.
2. ECOG PS 0-1
3. Be willing and able to provide written informed consent for the trial.
4. Be >= 18 years of age on day of signing informed consent.
5. Have measurable disease based on RECIST 1.1.
6. Demonstrate adequate organ function (as defined in Table 1 of the trial protocol) all screening tests should be performed within 10 days prior to confirmation of study eligibility.
7. Female patient of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to confirmation of study eligibility. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. For Concomitant cisplatin GFR>50ml/min, no contraindications to cisplatin (pre-existing tinnitus or neuropathy)

Exclusion Criteria:

1. Requires para-aortic radiotherapy
2. Has had previous pelvic radiotherapy
3. Has had bowel resection, history of inflammatory bowel disease or autoimmune condition
4. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
6. Has had a prior monoclonal antibody, chemotherapy, targeted small molecule therapy, or radiation therapy. Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
9. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 years from patients commencement
  To establish the maximum tolerated dose (MTD) of pembrolizumab that can be safely combined with radiotherapy, brachytherapy and cisplatin in the absence of dose limiting toxicities (DLTs)
Efficacy | 2 years from patients commencement
  Establish its efficacy on progression-free survival.

SECONDARY OUTCOMES:
Evaluate Toxicities of Treatment | Through study completion, up to 19 weeks after last dose of Pembrolizumab
  To evaluate acute toxicity as measured during treatment by CTCAE v4.0
Response Rates | 12 weeks (week 18), 6 months, 1 year and 2 following radiation treatment
  To determine response rates by RECIST v1.1
Presence / Absence of HPV | 12 weeks following radiation therapy (Week 18)
  To assess cervical HPV status using a cervical smear test for the presence / absence of HPV DNA/RNA.
Overall survival (OS) | Up to 2 years post treatment.
  To assess OS
Late Radiotherapy Toxicity | 12 weeks (study week 18), 6 months, 1 year and 2 years following radiation therapy
  To evaluate late radiotherapy toxicity as assessed by LENTSOM
Progression Free survival (PFS) | Up to 2 years post treatment.
  To assess PFS

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lalondrelle, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No